CLINICAL TRIAL: NCT01571245
Title: Predicting Treatment Response Using Psychophysiologic Reactivity Measures
Status: Completed | Type: Observational
Sponsor: Central Arkansas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 252121; PTRUPRM (Other: Central Arkansas Veterans Healthcare System)
Record Dates: First submitted 2012-03-27; First posted 2012-04-05 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Heart rate variability; Attentional Bias
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Veterans with PTSD: Operation Enduring Freedom/Operation Iraqi Freedom/Operation New Dawn (OEF/OIF/OND) veterans who are ages 18 to 60 and currently in or about to start treatment for deployment-related Post-Traumatic Stress Disorder (PTSD) at the Central Arkansas Veterans Healthcare System Mental Health Clinics.

SUMMARY:
Objective psychophysiologic reactivity data may be useful for predicting post-traumatic stress disorder (PTSD) treatment response. Given the variety of PTSD treatments and the lack of a clearly superior treatment, a reliable and valid approach to predicting treatment response is needed.

Specific Aims: 1). Evaluate the clinical utility of psychophysiologic reactivity measures to predict overall PTSD symptom response among OEF/OIF/OND (Operation Enduring Freedom/Operation Iraqi Freedom/Operation New Dawn) veterans receiving treatment for PTSD. 2). Evaluate the clinical utility of psychophysiologic reactivity measures to predict psychosocial functioning and health-related quality of life (HRQoL) response among OEF/OIF/OND veterans in treatment for PTSD. Exploratory). Develop psychophysiologic, neuropsychological, and/or self-report models to predict PTSD symptom response to pharmacotherapy, psychotherapy, and combined pharmacotherapy/psychotherapy. The investigators will divide psychophysiologic reactivity predictors into two groups: heart rate variability and attentional bias (eye gaze tracking and modified Stroop). The investigators will collect observational and longitudinal data from a treatment-seeking sample of 50 OEF/OIF/OND veterans with PTSD recruited from the Central Arkansas Veterans Healthcare System (CAVHS) Mental Health Clinics.

DETAILED DESCRIPTION:
All subjects will complete a baseline assessment including self-report data and psychophysiologic reactivity measures. Trained research assistants will collect psychophysiologic reactivity data. The investigators will collect the 3-month data in-person. At 6-months, self-report data will be collected in-person. If study participant is unable to complete the 6-month assessment in person the investigators will attempt to collect the self-report data by phone. The study instruments have all been previously administered by telephone. The project coordinator will schedule and track the participants using the telephone. The project coordinator will call participants to remind them about follow-up appointments. The consent form will also include the name and phone number of at least one contact person.

Psychophysiologic reactivity measures will be collected first to minimize fatigue. In addition, the psychophysiologic reactivity measures are context dependent and the investigators do not want the psychophysiologic measures to be primed by symptom reporting. Heart rate variability data will be collected at baseline for five minutes prior to other testing and then continued during eye gaze tracking and modified Stroop testing.

ELIGIBILITY:
Inclusion Criteria:

* OEF/OIF/OND Veterans
* Ages 18 to 60 (The investigators chose to limit the recruitment age to 60 because heart rate variability decreases dramatically with age and therefore may not demonstrate the variability necessary for use in a prediction model.)
* Currently in or about to start treatment for deployment-related PTSD at Mental Health Clinics
* PTSD symptom severity score using the PTSD Checklist-Civilian version of 40 or greater
* Able to provide the name and phone number of at least one contact person in case of difficulty locating participant for the follow-up assessment.

Exclusion Criteria:

* Current diagnosis of schizophrenia
* Daily use of benzodiazepines except as needed for sleep,
* Daily use of beta-blockers
* Plans to leave the area within 6 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Veterans receiving or seeking treatment at the Central Arkansas Veterans Healthcare Administration Mental Health Clinics.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2012-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in Eye-gaze Tracking | from Baseline to 6 months
  This measures attentional bias.

SECONDARY OUTCOMES:
Change in Modified Stroop | from Baseline to 6 months
  This measures attentional bias
Change in Heart rate variability | from Baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: John Spollen, MD, Principal Investigator — Central Arkansas Veterans Healthcare System
Locations (1):
- CAVHS Eugene Towbin VA Medical Center, North Little Rock, Arkansas, United States